CLINICAL TRIAL: NCT04381169
Title: Effect of Early Weight-based Aggressive Versus Non-aggressive Goal-directed Fluid Resuscitation in the Early Phase of Acute Pancreatitis: an Open-label Multicenter Randomized-controlled Trial
Brief Title: Aggressive Versus Non-aggressive Goal-directed Fluid Resuscitation in Acute Pancreatitis
Acronym: WATERFALL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Increased frequency of fluid overload on the aggressive fluid resuscitation arm of treatment
Sponsor: Enrique de-Madaria (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Asociación Española de Gastroenterología (Other); Asociación Española de Pancreatología (Unknown)
Responsible Party: Sponsor-Investigator, Enrique de-Madaria, Principal Investigator of the AUGH Clinical Pancreatology Research Group, Hospital General Universitario de Alicante
Organization: Hospital General Universitario de Alicante (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIM HGUA 2019/003; PI19/01628 (Other Grant/Funding Number: Instituto de Salud Carlos III); 2019-000788-26 (EudraCT Number)
Record Dates: First submitted 2020-05-02; First posted 2020-05-08 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; fluid resuscitation; therapy; outcomes; randomized controlled trial; Ringer lactate; Lactated Ringer's solution
MeSH Terms: conditions — Pancreatitis | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aggressive fluid resuscitation (Experimental): Lactated Ringer Solution 20 ml/kg bolus (administered over 2 hours) followed by an infusion of 3 ml/kg/h.
  At 12(±4) hours:
  A) Hypovolemia: same bolus and infusion B) No hypovolemia: infusion of lactated Ringer Solution 1.5 ml/kg/h C) Fluid overload: infusion rate of lactated Ringer Solution will be decreased or stopped
  Similar adjustments are repeated at 24(±4), 48(±4) and 72(±4) hours
  Fluid resuscitation is maintained at least 48h, and then it can be stopped in case of tolerating oral feeding for at least 8 hours
  Interventions: Drug: Lactated Ringer Solution
- Moderate fluid resuscitation (Experimental): At recruitment:
  A) Hypovolemia: Lactated Ringer Solution 10 ml/kg bolus (administered over 2 hours) followed by an infusion of 1.5 ml/kg/h.
  B) No hypovolemia: infusion of lactated Ringer Solution of 1.5 ml/kg/h (no bolus).
  At 12(±4) hours:
  A) Hypovolemia: same bolus and infusion B) No hypovolemia: infusion of lactated Ringer Solution 1.5 ml/kg/h C) Fluid overload: infusion rate of lactated Ringer Solution will be decreased or stopped
  Similar adjustments are repeated at 24(±4), 48(±4) and 72(±4) hours
  Fluid resuscitation can be stopped before the first 48h in case of tolerating oral feeding for at least 8 hours
  Interventions: Drug: Lactated Ringer Solution

INTERVENTIONS:
Drug: Lactated Ringer Solution — Comparison of aggressive versus moderate Lactated Ringer-based fluid resuscitation
  Other Names: Aggressive fluid resuscitation; Moderate fluid resuscitation; Restrictive fluid resuscitation

SUMMARY:
WATERFALL is an investigator-initiated international multicenter open-label randomized clinical trial comparing aggressive versus moderate fluid resuscitation in acute pancreatitis. The main outcome variable will be the proportion of patients with moderate-to-severe AP. Aggressive fluid resuscitation will consist in Lactated Ringer Solution (LR) 20 ml/kg bolus (administered over 2 hours) followed by LR 3 ml/kg/h and moderate a LR bolus 10 ml/kg in case of hypovolemia or no bolus in patients with normal volemia, followed by LR 1.5 ml/kg/h. The patients will be assessed at 3 (±1), 12 (±4), 24 (±4), 48 (±4) and 72 (±4) hours from recruitment, and fluid resuscitation will be adjusted to the patient´s clinical and analytical status according to a protocol. Subgroup analysis will include patients with systemic inflammatory response syndrome (SIRS) at admission, with persistent (>48h) SIRS and with hypovolemia at admission.

Based on available data (Sternby et al, Ann Surg 2019) we expect a 35% incidence of moderate to severe AP in the moderate arm. Sample sizes of 372 per arm of treatment (744 patients) achieve 80% power to detect a difference of 10% between the treatment arms at a significance level (alpha) of 0.05 using a two-sided z-testNA, assuming a 10% dropout. These results assume that 3 sequential tests are made using the O'Brien-Fleming spending function to determine the test boundaries.

All analyses will be performed on an intention-to-treat basis. The trial could be stop early for efficacy (primary end-point) if the observed two-sided P value is <0.0002 at the first interim analysis (after 1/3 of patients have been enrolled) or is <0.012 at second interim analysis (after 2/3 of patients have been enrolled), favoring aggressive fluid resuscitation. At final analysis, the hypothesis that the incidence of moderate-to-severe pancreatitis is similar in the two treatment arms will be rejected if p<0.046

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater or equal to 18 presenting to one of the collaborating centers
* Diagnosis of acute pancreatitis according to the revised Atlanta classification which requires 2 of the following 3 criteria: A) Typical abdominal pain; B) Increase in serum amylase or lipase levels higher than 3 times the upper limit of normality; and C) Signs of AP in imaging.

Exclusion Criteria:

* Uncontrolled arterial hypertension (systolic blood pressure >180 and/or diastolic blood pressure 100 mmHg);
* New York Heart Association Class II hear failure (slight limitation of physical activity; fatigue, palpitations or dyspnea with ordinal physical activity) or worse, or ejection fraction<50% in the last echocardiography;
* Decompensated cirrhosis (Child's Class B or C);
* Hyper or hyponatremia (<135 or >145 mEq/l);
* Hyperkalemia (>5 mEq/l);
* Hypercalcemia (albumin or protein-corrected calcium>10.5 mg/dl);
* Chronic kidney failure (basal glomerular filtration rate <60 mL/min/1.73m2);
* Clinical signs or symptoms of volume overload or heart failure at recruitment (dyspnea, peripheral edema, pulmonary rales, or evident increased jugular ingurgitation at 45º);
* Shock or respiratory failure according to the revised Atlanta classification at recruitment (non-fluid responding systolic blood pressure< 90 mmHg, PaO2/FIO2≤300 mmHg);
* Time from pain onset to arrival to emergency room >24h;
* Time from confirmation of pancreatitis to randomization >8h;
* Severe comorbidity associated with an estimated life expectancy <1 year;
* Confirmed chronic pancreatitis (in case of recurrent alcoholic pancreatitis a recent (<6 months) CT scan/MRI or endoscopic ultrasound is needed to rule out chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Moderate-to-severe acute pancreatitis | From admission to discharge, up to 24 weeks
  Moderate or severe category of the Revised Atlanta Classification (Banks et al, Gut 2013)

SECONDARY OUTCOMES:
Death and/or persistent organ failure and/or infection of pancreatic necrosis | From admission to discharge, up to 24 weeks
  Analyzed as a composite endpoint and each of its components, includes in-hospital mortality, persistent organ failure (according to the revised Atlanta classification, Banks et al, Gut 2013) or infection of pancreatic necrosis
Fluid overload | From admission to discharge, up to 24 weeks
  Fluid overload is defined by the absence of Acute Respiratory Distress Syndrome and at least 2 of the following 3 criteria (based on Sharma et al, Lancet Diabetes Endocrinol 2016, with modifications):
  Criteria 1. Hemodynamic-imaging evidence (≥1):
  * Non-invasive diagnostic evidence of heart failure (i.e., echocardiographic, cardiac MRI)
  * Radiographic evidence of pulmonary congestion
  * Invasive cardiac catheterization suggesting evidence of heart failure (i.e., pulmonary capillary wedge pressure [or left ventricular end-diastolic pressure] >18 mm Hg, right arterial pressure [or central venous pressure] >12 mm Hg, or cardiac index < 2·2 L/min per m2)
  Criteria 2. Heart failure symptoms (1):
  - Dyspnea
  Criteria 3. Heart failure signs (≥1):
  * Peripheral edema
  * Pulmonary rales or crackles, or crepitation
  * Increased jugular venous pressure, hepatojugular reflux, or both
Shock | From admission to discharge, up to 24 weeks
  Systolic blood pressure <90 mmHg after fluid resuscitation
Respiratory failure | From admission to discharge, up to 24 weeks
  PaO2/FIO2<300
Kidney failure | From admission to discharge, up to 24 weeks
  Creatinine >1.9 mg/dL
Local complications (acute peripancreatic fluid collections/ pancreatic necrosis/peripancreatic necrosis) | From admission to discharge, up to 24 weeks
  As described on the revised Atlanta classification, Banks et al, Gut 2013
Length of hospital stay | From admission to discharge, up to 24 weeks
Intensive care unit stay | From admission to discharge, up to 24 weeks
  Need for intensive care unit (ICU) admission, and days admitted in the ICU
Need for invasive treatment | From admission to discharge, up to 24 weeks
  Endoscopic, percutaneous or surgical treatment of acute pancreatitis complications
Need for nutritional support | From admission to discharge, up to 24 weeks
  Need for enteral/parenteral feeding
PAN-PROMISE scale | At 12, 24, 48 and 72 hours
  Score on an acute pancreatitis Patient-Reported Outcome Measurement
C-reactive protein | 48 and 72 hours
  Blood levels of C-reactive protein
Systemic inflammatory response syndrome (SIRS) | Baseline, 12, 24, 48 and 72 hours
  SIRS at the different checkpoints. Presence of persistent (>48h) SIRS

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Alicante, Alicante
  - Hospital General Universitario de Alicante, Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Derived] de-Madaria E, Buxbaum JL, Maisonneuve P, Garcia Garcia de Paredes A, Zapater P, Guilabert L, Vaillo-Rocamora A, Rodriguez-Gandia MA, Donate-Ortega J, Lozada-Hernandez EE, Collazo Moreno AJR, Lira-Aguilar A, Llovet LP, Mehta R, Tandel R, Navarro P, Sanchez-Pardo AM, Sanchez-Marin C, Cobreros M, Fernandez-Cabrera I, Casals-Seoane F, Casas Deza D, Lauret-Brana E, Marti-Marques E, Camacho-Montano LM, Ubieto V, Ganuza M, Bolado F; ERICA Consortium. Aggressive or Moderate Fluid Resuscitation in Acute Pancreatitis. N Engl J Med. 2022 Sep 15;387(11):989-1000. doi: 10.1056/NEJMoa2202884. PMID 36103415

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04381169/Prot_SAP_000.pdf